CLINICAL TRIAL: NCT03764332
Title: Evaluation of the Static Stability of Footwear: A Clinical Trial
Brief Title: Evaluation of the Static Stability of Footwear
Acronym: EEECS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JOSE MANUEL SANCHEZ SAEZ (Other)
Responsible Party: Sponsor-Investigator, JOSE MANUEL SANCHEZ SAEZ, Principal investigator, Universidade da Coruña
Organization: Universidade da Coruña (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1402201803718
Record Dates: First submitted 2018-11-27; First posted 2018-12-05 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Postural; Strain
Keywords: Footwear; Barefoot
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stabilometry (Other): The Podoprint pressure platform was used as a measuring device. The Podoprint platform is a low profile floor platform consisting of 1.4 sensors / cm2 with a sampling frequency of 40Hz.
  Interventions: Device: Stabilometry

INTERVENTIONS:
Device: Stabilometry — To evaluate the static balance of subjects when barefoot and when using three types of footwear with their eyes closed or open.
  Other Names: Eyes open and eyes closed

SUMMARY:
Introduction: Postural control is a crucial factor for maintaining balance while standing and walking. The shoe has a role to play in postural stability.

Objectives: To evaluate the static balance of subjects when barefoot and when using three types of footwear with their eyes closed or open.

Material and methods:

DETAILED DESCRIPTION:
Each participant was asked to focus on a white mark 2 cm in diameter, positioned on a screen 2 m in front of them at eye level. This was done to standardize the data collection and minimize any variation in postural stability caused by changes in the visual field. Each participant was asked to remain in this position for a period of 30 seconds, while the data was collected. Three repetitions were made for each condition to obtain an average value. The condition on footwear and open / closed eyes was randomized to reduce the learning effect. On the other hand to reduce fatigue, each participant was allowed to rest for 5 minutes between shoe changes.

The size of the sample was calculated with the software of the Clinical Epidemiology and Biostatistics Unit. Complexo Hospitalario Universitario de A Coruña. University of A Coruña (www.fisterra.com). The estimated sample size estimated was calculated to be at least 16 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance and signature of informed consent.
* Persons aged between 25-35 years.
* People with a weight between 40 and 95kg.
* People with a height between 1.50 and 1.90m

Exclusion Criteria:

* People with surgical history of lower limbs.
* People with systemic pathology / algia that can alter the physiological static pattern.
* Congenital deformities or acquired in childhood.
* If after a complete exploration in decubitus, sitting, static standing and gait dynamics, any anomaly that could negatively influence the acquisition of data for the study was detected.
* Patients who do not accept or sign the informed consent

Ages: 25 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-04 (Actual)

PRIMARY OUTCOMES:
Stroke length | 30 seconds
  Length traveled by the pressure center (CoP), forming a line called oscillatory ball. In mm. The Podoprint pressure platform was used as a measuring device.
  Quantitative variable
Stroke surface | 30 seconds
  Area of the smallest ellipse able to encompass the oscillating ball. In mm. The Podoprint pressure platform was used as a measuring device.
  Quantitative variable
Relationship between Length / surface | 30 seconds
  Value resulting from the relationship between the two previous measures. The Podoprint pressure platform was used as a measuring device.
  Quantitative variable
Average swing speed | 30 seconds
  Average speed that reaches the displacement of the center of pressures. The Podoprint pressure platform was used as a measuring device.
  Quantitative variable
Lateral velocity | 30 seconds
  Average speed of oscillation in its axis of ordinates. The Podoprint pressure platform was used as a measuring device. Quantitative variable
Forward speed | 30 seconds
  Average oscillation speed on its abscissa axis. The Podoprint pressure platform was used as a measuring device. Quantitative variable
Average displacement in the X axis | 30 seconds
  Average of the displacements made by the center of pressures in the axis of ordinates. The Podoprint pressure platform was used as a measuring device.
  Quantitative variable
Average displacement on the Y axis | 30 seconds
  Average of the displacements made by the center of pressures on the abscissa axis. The Podoprint pressure platform was used as a measuring device.
  Quantitative variable

CONTACTS AND LOCATIONS:
Overall Officials: Jose Sanchez Saez, Podólogo, Principal Investigator — Universidade da Coruña
Locations (1):
- Clínica López del Amo, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanchez-Saez JM, Palomo-Lopez P, Becerro-de-Bengoa-Vallejo R, Calvo-Lobo C, Losa-Iglesias ME, Lopez-Del-Amo-Lorente A, Lopez-Lopez D. Stability of Three Different Sanitary Shoes on Healthcare Workers: A Cross-Sectional Study. Int J Environ Res Public Health. 2019 Jun 16;16(12):2126. doi: 10.3390/ijerph16122126. PMID 31208123